CLINICAL TRIAL: NCT07307235
Title: Efficacy and Safety of iGlarLixi Versus Standard of Care in a Real-world Adult China Population With Uncontrolled Type 2 Diabetes on Oral Agents-a Pragmatic Randomized Controlled Trial
Brief Title: Efficacy and Safety of iGlarLixi Versus Standard of Care in a Real-world Adult China Population With Uncontrolled Type 2 Diabetes on Oral Agents
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Sanofi (China) Investment Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250424044409703
Record Dates: First submitted 2025-11-28; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; iGlarLixi; RCT
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine; lixisenatide; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iGlarLixi group (Experimental): The investigational drug is iGlarLixi. Participants will receive subcutaneous injections of iGlarLixi with the OAD treatment regimen being appropriately maintained or adjusted as intensification therapy in routine clinical practice.
  Interventions: Drug: iGlarLixi (insulin glargine/lixisenatide)
- Standard of care (SOC) group. (Active Comparator): The control drug treatment is standard of care (basal insulin or premixed insulin, excluding any GLP-1 receptor agonist-containing drugs). Participants will receive standard of care with the OAD treatment regimen being maintained or appropriately adjusted as an intensification treatment during routine clinical practice.
  Interventions: Drug: standard of care (basal insulin or premixed insulin, excluding any GLP-1 receptor agonist-containing drugs)

INTERVENTIONS:
Drug: iGlarLixi (insulin glargine/lixisenatide) — The investigational drug is iGlarLixi. Participants will receive subcutaneous injections of iGlarLixi with the OAD treatment regimen being appropriately maintained or adjusted as intensification therapy in routine clinical practice.
  Arms: iGlarLixi group
Drug: standard of care (basal insulin or premixed insulin, excluding any GLP-1 receptor agonist-containing drugs) — The control drug treatment is standard of care (basal insulin or premixed insulin, excluding any GLP-1 receptor agonist-containing drugs). Participants will receive standard of care with the OAD treatment regimen being maintained or appropriately adjusted as an intensification treatment during routine clinical practice.
  Arms: Standard of care (SOC) group.

SUMMARY:
This study is a prospective, open-label, multicenter, parallel-group, positive-controlled, and pragmatic randomized clinical trial (pRCT). It will compare the efficacy and safety of iGlarLixi versus standard of care in adult T2DM patients with poor glycemic control, who are using 1 to 3 OADs in a real-world clinical practice setting. A total of 1,316 subjects from approximately 40 research centers in China will be randomly assigned in a 1:1 ratio to one of the following treatment groups: Group 1: iGlarLixi for blood glucose control; and Group 2: Standard of care for diabetes (basal insulin or premixed insulin, excluding any GLP-1RA-containing drugs). Considering the substantial difference in intervention methods between the two groups, the study is designed as non-blinded with an open-label approach.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 of age inclusive, at the time of signing the informed consent.
2. Type 2 diabetes mellitus diagnosis.
3. Participants who are treated for at least 3 months prior to the screening visit with an adequate dose of 1-3 OADs (Met, SGLT2i, alpha-GI, glinide or SU).
4. HbA1c 7.5-11%
5. Further intensification with an additional antidiabetic injectable medication is indicated to achieve glycaemic target at the discretion of the study physician according to approval labelling.

Participants who have signed informed consent form (ICF).

Exclusion Criteria:

1. Diagnosed with T1DM
2. BMI <20 kg/m2 or BMI ≥40 kg/m2
3. Treatment with more than 3 oral antidiabetic medications, or any injectable medication in a period of 30 days before the day of eligibility assessment. Temporary/emergency use of insulin is allowed, as is prior insulin treatment for gestational diabetes.
4. Contraindications to iGlarLixi according to the China NMPA approved label.
5. Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening, or any major systemic disease resulting in short life expectancy that in the opinion of the Investigator would restrict or limit the patient's successful participation for the duration of the study.
6. Participants who involved in other clinical trial within 3 months prior to the time of screening visit.
7. Participant who has a severe renal function impairment with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2
8. Pregnant or breast-feeding woman.
9. Woman of childbearing potential not protected by highly effective contraceptive method of birth control and/or who is unwilling or unable to be tested for pregnancy.
10. Conditions/situations such as:

Participant with short life expectancy. Participant with conditions/concomitant diseases making him/her not evaluable for the primary efficacy endpoint (eg, hemoglobinopathy or hemolytic anemia, receipt of blood or plasma products within 3 months prior to screening).

Participant with conditions/concomitant diseases precluding his/her safe participation in this study (eg, active malignant tumor, major systemic diseases, presence of clinically significant diabetic retinopathy or presence of macular edema likely to require laser treatment within the study period).

Uncooperative or any condition that could make the participant potentially non-compliant to the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1316 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
hemoglobin A1c (HbA1c) change | from baseline to week 24
  The primary endpoint is the change in HbA1c from baseline to week 24 (percentage [%]).

SECONDARY OUTCOMES:
Proportion of subjects achieving HbA1c < 7% at week 24 | 24 weeks
Proportion of subjects achieving HbA1c < 7%, with no weight gain and no hypoglycemia (defined as ADA grades 1, 2, or 3) at week 24 | 24 weeks
Change in weight from baseline to week 24 | 24 weeks
Change in Fasting plasma glucose from baseline to Week 24. | 24 weeks
Change in 7-point self-monitored plasma glucose (SMPG) profile from baseline to Week 24 (each time point and average daily value). | 24 weeks
Proportion of participants reaching HbA1c target <7% with no hypoglycemia (defined as ADA level 1, 2 or 3) at Week 24. | 24 weeks
Proportion of participants reaching HbA1c target <7% with no clinically relevant hypoglycemia (defined as ADA level 2 or 3) at Week 24 | 24 weeks
Change in CGM metrics(TIR / TAR / TBR /mean daily glucose / TITR / CV / GMI / SD of mean glucose) from baseline to Week 24 | 24 weeks
Change in proportion of patients achieving CGM metrics targets (TIR / TAR / TBR / TITR / CV) from baseline to Week 24 | 24 weeks
Change in waist from baseline to Week 24 | 24 weeks
Total insulin dose in each group at Week 24 | 24 weeks
Change in fasting C-peptide from baseline to Week 24 | 24 weeks
Percentage of participants requiring rescue therapy during the 24-week treatment period | 24 weeks
Time to first study drug discontinuation during 24 weeks (day) | 24 weeks
Time to first treatment intensification (add-on) or change (switch) after randomization during 24 weeks (day) | 24 weeks
Study drug medication adherence of the study, as measured by medication possession ratio (MPR) (%) | 24 weeks
Change from baseline to Week 24 in diabetes medication treatment satisfaction scores (total score and by sub scales), using the treatment related impact measure diabetes (TRIM-D) questionnaire. | 24 weeks
  TRIM scores range from 0 to 100 with a higher score indicating a better health state.
All cause healthcare resource utilization (HCRU) from baseline to EOT（end of treatment | 24 weeks
Incidence and event rate of hypoglycemia | 24 weeks
  any hypoglycemia, ADA grades 1-2-3
Incidence and event rate of Adverse events (AE) | 24 weeks
Incidence and event rate of serious adverse events (SAE) | 24 weeks
  An SAE is defined as any adverse event occurring at any dose that meets one or more of the following criteria:
  1. Results in death
  2. Is life-threatening
  3. Requires hospitalization or prolongs existing hospitalization
  4. Results in persistent or significant disability/incapacity
  5. Is a congenital anomaly/birth defect
  6. Other important medical events
Incidence and event rate of adverse events of special interest (AESI) | 24 weeks
  The following events are designated as AESIs:
  1. Pregnancy in female subjects or pregnancy in female partners of male subjects exposed to IMP/NIMP
  2. Symptomatic overdose of IMP/NIMP (serious or non-serious)
  3. Alanine aminotransferase (ALT) elevation >3×ULN
Incidence and event rate of AEs leading to treatment discontinuation, vital signs, and safety laboratory test values. | 24 weeks

OTHER OUTCOMES:
Change in CRP from baseline to week 24. | from baseline to week 24
  Change in CRP from baseline to week 24.